CLINICAL TRIAL: NCT02631447
Title: A Three Arms Prospective, Randomized Phase II Study to Evaluate the Best Sequential Approach With Combo Immunotherapy (Ipilimumab/Nivolumab) and Combo Target Therapy (LGX818/MEK162) in Patients With Metastatic Melanoma and BRAF Mutation
Brief Title: Sequential Combo Immuno and Target Therapy (SECOMBIT) Study
Acronym: SECOMBIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Melanoma Onlus (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECOMBIT; 2014-004842-92 (EudraCT Number)
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; BRAF mutation
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Combo Target/Combo Immuno (Experimental): Combo Target (LGX818 450 mg p.o. od + MEK162 45 mg p.o. bid) until PD; then Combo Immuno (nivolumab 1 mg/kg solution IV combined with ipilimumab 3 mg/kg solution IV every 3 weeks for 4 doses then nivolumab 3 mg/kg solution IV every 2 weeks) until PD
  Interventions: Drug: LGX818; Drug: MEK162; Drug: Nivolumab; Drug: Ipilimumab
- Arm B: Como immuno/Combo Target (Experimental): Combo Immuno (nivolumab 1 mg/kg solution IV combined with ipilimumab 3 mg/kg solution IV every 3 weeks for 4 doses then nivolumab 3 mg/kg solution IV every 2 weeks) until PD; then Combo Target (LGX818 450 mg p.o. od + MEK162 45 mg p.o. bid) until PD
  Interventions: Drug: LGX818; Drug: MEK162; Drug: Nivolumab; Drug: Ipilimumab
- Arm C: Sandwich (Experimental): Combo Target (LGX818 450 mg p.o. od + MEK162 45 mg p.o. bid) for 8 weeks followed by Combo Immuno (nivolumab 1 mg/kg solution IV combined with ipilimumab 3 mg/kg solution IV every 3 weeks for 4 doses then nivolumab 3 mg/kg solution IV every 2 weeks) until PD; then Combo Target (LGX818 450 mg p.o. od + MEK162 45 mg p.o. bid) until PD
  Interventions: Drug: LGX818; Drug: MEK162; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: LGX818 — LGX818 450 mg p.o. od
  Other Names: Combo target; IMP3
Drug: MEK162 — MEK162 45 mg p.o. bid
  Other Names: Combo target; IMP4
Drug: Nivolumab — Nivolumab 1 mg/kg solution IV combined with ipilimumab 3 mg/kg solution IV every 3 weeks for 4 doses then nivolumab 3 mg/kg solution IV every 2 weeks
  Other Names: Combo Immuno; IMP1
Drug: Ipilimumab — Nivolumab 1 mg/kg solution IV combined with ipilimumab 3 mg/kg solution IV every 3 weeks for 4 doses then nivolumab 3 mg/kg solution IV every 2 weeks
  Other Names: Combo Immuno; IMP2

SUMMARY:
To evaluate the best sequencing approach with the combination of target agents (LGX818 plus MEK162) and the combination of immunomodulatory antibodies (ipilimumab plus nivolumab) in patients with metastatic melanoma and BRAF V600 mutation.

DETAILED DESCRIPTION:
The combination BRAF (B-raf murine sarcoma viral oncogene homolog B1) inhibitor plus mitogen-activated protein kinase (MEK) inhibitor seems to be more effective in the V600 BRAF mutated advanced melanoma patients compared to treatment with the BRAF inhibitors alone. In fact, a phase I-II study showed a better overall response rate (ORR) and progression-free survival (PFS) in the combination arm (dabrafenib plus trametinib) respect to the single agent treatment (dabrafenib): 76% and 9.4 months versus 54% and 5.8 months respectively. Another phase I study with a similar combination (vemurafenib plus cobimetinib) showed an ORR of 85% in vemurafenib-naïve patients.

Recently, the results of a phase I study about the combination ipilimumab plus nivolumab have been reported. In this study at the selected schedule (ipilimumab 3 mg/kg and nivolumab 1 mg/kg), 53% of patients had an objective response, all with tumor reduction of 80% or more. Reponses were durable, although longer follow-up is needed.

A recent phase I study has shown a high rate of liver toxicity with the combo ipilimumab plus vemurafenib . which makes difficult a combination with these two different drugs. Moreover, a better efficacy of the sequencing treatment BRAF inhibitors/ipilimumab vs. the single agent treatment was also observed; for this reason it was also suggested to start immunotherapy treatment in the BRAF V600 mutated melanoma population as first option, in order to increase the percentage of patients who can benefit from the sequencing, considering the possibility of a fast progression of the disease after the BRAF inhibitors treatment.

Taking into account these considerations, it seems impossible to think to combine all the four compounds (the target agents and immunomodulating monoclonal antibodies). The risk of a high rate of toxicity is realistic and would render this approach inapplicable.

Sequencing with these different combinations seems to be more feasible. However, also in this case it would be important to start with the best combination in order to give to the patients the best chance to increase the overall survival.

The aim of this prospective randomized phase II study is to evaluate the sequencing of these two different combinations and evaluate which is the best of these approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥ 18 years;
2. Histologically confirmed stage III (unresectable) or stage IV melanoma with the BRAF V600 mutation. Patients with mucosal melanoma (but not those with ocular melanoma) are eligible for study participation;
3. Treatment naïve for metastatic disease patients. Previous adjuvant treatment, included checkpoint inhibitors anti CTLA-4, anti PD-1/PDL-1 is allowed, except for stage IV (if completed at least 6 weeks prior to randomization, and all related adverse events have either returned to baseline or stabilized). BRAF inhibitor treatment in adjuvant setting is not permitted.
4. Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria;
5. Presence of BRAF V600E or V600K mutation in tumor tissue prior to enrollment;
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1;
7. Tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses. An archive sample is mandatory at the screening visit; however, a new sample collection would be preferable;
8. Female subjects of childbearing potential must have a negative pregnancy test result at baseline and must practice two highly effective methods of contraception for the total study duration plus 23 weeks (i.e. 30 days plus the time required for nivolumab to undergo five half lives) after the last dose of nivolumab and ipilimumab and 30 days after the last dose of binimetinib and encorafenib for female subjects. Additional pregnancy testing must be performed every 6 weeks during the treatment Combo-Immuno and every 4 weeks during the treatment Combo-Target, as well as at the end of the systemic exposure;
9. Men who are sexually active with women of childbearing potential must practice a reliable method of contraception for the total study duration plus 31 weeks (i.e. 80 days plus the time required for nivolumab to undergo five half lives) after the last dose of nivolumab and ipilimumab and 90 days after the last dose of binimetinib and encorafenib;
10. Adequate bone marrow haematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L AND platelet count ≥ 100 x 109/L AND haemoglobin ≥ 9 g/dL;
11. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) AND aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 X ULN (< 5 x ULN if liver metastases);
12. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥ 50 mL/min in females (calculated according to Cockroft-Gault formula);
13. Serum calcium levels, international normalised ratio (INR) and partial thromboplastin time were within normal limits;
14. Life expectancy of at least 3 months;
15. Ability to understand study-related patient information and provision of written informed consent for participation in the study.
16. Adequate electrolytes at Baseline, defined as serum potassium and magnesium levels within institutional normal limits (Note: replacement treatment to achieve adequate electrolytes will be allowed).
17. Adequate cardiac function:

    * left ventricular ejection fraction (LVEF) ≥ 50% as determined by a multigated --acquisition (MUGA) scan or echocardiogram,
    * QTc interval ≤ 480 ms (preferably the mean from triplicate ECGs)

Exclusion Criteria:

1. Active brain metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration;
2. Subjects with active, known or suspected autoimmune disease;
3. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment;
4. Prior treatment for stage III (unresectable) or stage IV melanoma with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) antibody;
5. Female subjects who are pregnant (positive pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control;
6. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study;
7. Patients with a history of uncontrolled cardiovascular or interstitial lung disease and evidence or risk of retinal vein occlusion or central serous retinopathy (patients with a history of cardiovascular or interstitial lung disease and evidence or risk of retinal vein occlusion or central serous retinopathy (past or present evidence of rethinophaty central serous retinopathy - CSR -, occlusion of retinal - RVOo retinal degenerative disease) or ophthalmopathy, which according to the ophthalmologic evaluation at baseline could be considered a risk factor for CSR / RVO ( eg. cupping of the optic disc, visual field defect, intraocular pressure - (eg: central IOP - > 21 mmHg);
8. Previous or concurrent malignancy. Exceptions: adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to study entry; or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry
9. History of Gilbert's syndrome;
10. Inability to regularly access centre facilities for logistical or other reasons;
11. History of poor co-operation, non-compliance with medical treatment, or unreliability;
12. Participation in any interventional drug or medical device study within 30 days prior to treatment start.
13. Positive test for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
14. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
15. Receipt of live vaccine within 30 days prior to study drug administration.
16. History of severe or life-threatening skin adverse events or reactions to drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 24 month
  OS is defined as the time between the date of randomization and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive. OS data will be collected continuously while subjects are on study medication and every 3 months via in-person or phone contact after discontinuation of study medication

SECONDARY OUTCOMES:
Total Progression free survival | Baseline (Day 1), every 6 weeks until second disease progression is documented (Approximately around 2 years)
  PFS is defined as the time between the date of randomization and the first date of documented progression, as determined by the investigator, or death due to any cause, whichever occurs first.
  Tumor responses will be assessed by the Investigator according to RECIST Criteria (version 1.1)
Percentage of patients alive at 2 and 3 years; | Time Frame: at 24^ and 36^ month
  Percentage of patients alive at 2 and 3 years will be reported using Wilson score intervals.
Best overall response rate (BORR); | Time Frame: up to 24 months
  It will be calculated as the percentage of ITT population patients who have a CR o o PR before any evidence of progression (as defined by RECIST).
Duration of response (DoR); | Time Frame: up to 24 months
  It will be calculated as the percentage of ITT population patients who have a CR o o PR before any evidence of progression (as defined by RECIST).
Toxicity of the investigational medicinal products (IMPs). | Time Frame: up to 24 months
  Safety and tolerability will be assessed in terms od AEs, laboratory data, ECG data, vitals signs and weight, which will be collected for all patients. AEs (both in terms od MedDRA preferred terms and CTCAE grade), laboratory data, ECG data, vital signs and weight will be listes individually by patient and summarized by treatment received. ECG changes will be summarized for each treatment group.
Quality of life and general health | Time Frame: up to 24 months
  Changes from baseline in EQ-5D and QLQ-C30 total score will be summarized by means of descriptive statistical methods.
3 years PFS rate | Time Frame: up to 36 months
  3 years PFS rate; calculated from the date of randomization;

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Ascierto, MD, Study Chair — Fondazione Melanoma Onlus
Locations (30):
- Austria (4):
  - Paracelsus Medical University, Salzburg, AT
  - Karl Landsteiner University of Health Sciencies - University Clinic, Sankt Pölten, AT
  - Medical University of Graz, Graz, AU
  - Medical University of Vienna, Vienna
- Hôpitaux Universitaires Saint-Louis, Paris, France
- University of Tuebingen, Tübingen, Germany
- University of Athens, Athens, Greece
- Italy (15):
  - IRCCS - Istituto Scientifico Romagnolo per la Cura e lo Studio dei Tumori (I.R.S.T) S.r.l., Meldola, Forlì-Cesena
  - National Institute of Cancer, Bari
  - Università degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - IRCCS San Martino - IST, Genova
  - Fondazione I.R.C.C.S. Istituto Nazionale dei Tumori, Milan
  - IEO - Istituto Europeo di Oncologia - IRCCS, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Giovanni Pascale", Naples
  - Azienda Ospedaliero Universitaria Federico II, Naples
  - Istituto Oncologico Veneto, Padua
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Dermopatico dell'Immacolata - IDI - IRCCS, Roma
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria - Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata di Udine, Udine
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, PL, Poland
- Spain (3):
  - Hospital Universitario Quiròn Dexeus, Barcelona, SP
  - Hospital Clínic Barcelona, Barcelona
  - Clinica Universidad de Navarra, Pamplona
- Karolinska University Hospital, Stockholm, Sweden
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ascierto PA, Mandala M, Ferrucci PF, Guidoboni M, Rutkowski P, Ferraresi V, Arance A, Guida M, Maiello E, Gogas H, Richtig E, Quaglino P, Lebbe C, Helgadottir H, Queirolo P, Spagnolo F, Tucci M, Del Vecchio M, Gonzalez-Cao M, Minisini AM, De Placido S, Sanmamed MF, Casula M, Bulgarelli J, Pisano M, Piccinini C, Piccin L, Cossu A, Mallardo D, Paone M, Vitale MG, Melero I, Grimaldi AM, Giannarelli D, Palmieri G, Dummer R, Sileni VC. Sequencing of Checkpoint or BRAF/MEK Inhibitors on Brain Metastases in Melanoma. NEJM Evid. 2024 Oct;3(10):EVIDoa2400087. doi: 10.1056/EVIDoa2400087. Epub 2024 Sep 24. PMID 39315864
- [Derived] Ascierto PA, Casula M, Bulgarelli J, Pisano M, Piccinini C, Piccin L, Cossu A, Mandala M, Ferrucci PF, Guidoboni M, Rutkowski P, Ferraresi V, Arance A, Guida M, Maiello E, Gogas H, Richtig E, Fierro MT, Lebbe C, Helgadottir H, Queirolo P, Spagnolo F, Tucci M, Del Vecchio M, Cao MG, Minisini AM, De Placido S, Sanmamed MF, Mallardo D, Paone M, Vitale MG, Melero I, Grimaldi AM, Giannarelli D, Dummer R, Sileni VC, Palmieri G. Sequential immunotherapy and targeted therapy for metastatic BRAF V600 mutated melanoma: 4-year survival and biomarkers evaluation from the phase II SECOMBIT trial. Nat Commun. 2024 Jan 2;15(1):146. doi: 10.1038/s41467-023-44475-6. PMID 38167503
- [Derived] Ascierto PA, Mandala M, Ferrucci PF, Guidoboni M, Rutkowski P, Ferraresi V, Arance A, Guida M, Maiello E, Gogas H, Richtig E, Fierro MT, Lebbe C, Helgadottir H, Queirolo P, Spagnolo F, Tucci M, Del Vecchio M, Gonzales Cao M, Minisini AM, De Placido S, Sanmamed MF, Mallardo D, Curvietto M, Melero I, Palmieri G, Grimaldi AM, Giannarelli D, Dummer R, Chiarion Sileni V. Sequencing of Ipilimumab Plus Nivolumab and Encorafenib Plus Binimetinib for Untreated BRAF-Mutated Metastatic Melanoma (SECOMBIT): A Randomized, Three-Arm, Open-Label Phase II Trial. J Clin Oncol. 2023 Jan 10;41(2):212-221. doi: 10.1200/JCO.21.02961. Epub 2022 Sep 1. PMID 36049147